CLINICAL TRIAL: NCT03289702
Title: A Randomized, Double-blind, Active Drug Controlled, Multi-Center, Phase I/III Clinical Trial to Evaluate the Efficacy and Safety of CORETOX® in Treatment of Post Stroke Upper Limb Spasticity
Brief Title: CORETOX® in Treatment of Post Stroke Upper Limb Spasticity (Phase3)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medy-Tox (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MT03-KR16MST907 (Phase3)
Record Dates: First submitted 2017-09-19; First posted 2017-09-21 (Actual); Last update posted 2021-12-07 (Actual); Status verified 2021-12

CONDITIONS: Muscle Spasticity
MeSH Terms: conditions — Muscle Spasticity | interventions — coretox; Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CORETOX® (Experimental)
  Interventions: Drug: CORETOX®
- BOTOX® (Active Comparator)
  Interventions: Drug: BOTOX®

INTERVENTIONS:
Drug: CORETOX® — Upper limb will be injected and evaluated in the study. Maximum injection dose is 360U.
  Arms: CORETOX®
Drug: BOTOX® — Upper limb will be injected and evaluated in the study. Maximum injection dose is 360U.
  Arms: BOTOX®

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of CORETOX® in the treatment of post-stroke upper limb spasticity

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients ≥ 19 years
* ≥ 6 months since the last stroke
* ≥ 2 points in the focal spasticity of wrist flexor and ≥ 1 point at least one of elbow flexor and finger flexor as measured on MAS(0 to 4)
* Informed consent has been obtained

Exclusion Criteria:

* Neuromuscular disorders such as Lambert-Eaton syndrome, myasthenia gravis, or amyotrophic lateral sclerosis
* History(within 4 months of screening visit) or planned(during study period) treatment with phenol or alcohol injection or surgery in the target limb
* History(within 4 months of screening visit) or planned(during study period) treatment with tendon lengthening in the target limb
* Fixed joint/muscle contracture
* Severe atrophy
* Concurrent treatment with an intrathecal baclofen
* Patients who have bleeding tendency or taking anti-coagulant
* Dysphagia and Breathing Difficulties
* History(within 4 months of screening visit) Planned(during study period) treatment with Botulinum Toxin
* Known allergy or sensitivity to study medication or its components
* Concurrent or planed Muscle relaxants and/or benzodiazepine medication If patient has taken these medication stable from one month before screening and no treatment changes are not planned during the study, participation is allowed.
* Current Physical, occupational, Splinting therapy These therapy regimens will be permitted if they have been stable in the one month before screening; no treatment and no changes are planned during the study.
* Patient who are participating in other clinical trials at the screening
* Females who are pregnant, breastfeeding, or planning a pregnancy during the study period, or female of childbearing potential, not using a reliable means of contraception.
* Patients who are not eligible for this study at the discretion of the investigator.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2017-11-13 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-11-09 (Actual)

PRIMARY OUTCOMES:
MAS(Modified Ashworth Scale)of wrist flexor | 4 weeks
  Change from baseline at week 4 for wrist flexor muscle tone as measured on the MAS(Modified Ashworth Scale)

SECONDARY OUTCOMES:
MAS(modified Ashworth Score)of elbow and finger flexor | 4 weeks after injection
  Change from baseline at week 4 for elbow flexor and finger flexor muscle tone as measured on MAS
MAS(modified Ashworth Score)of wrist, elbow and finger flexor | 8, 12 weeks after injection
  Change from baseline at week 8, 12 for wrist flexor, elbow flexor and finger flexor muscle tone as measured on MAS
Percentage of treatment responder at week 4, 8, 12 after injection | 4, 8, 12 weeks after injection
  A treatment response is defined as 1-point improvement on the MAS of injection site

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lee J, Chun MH, Ko YJ, Lee SU, Kim DY, Paik NJ, Kwon BS, Park YG. Efficacy and Safety of MT10107 (Coretox) in Poststroke Upper Limb Spasticity Treatment: A Randomized, Double-Blind, Active Drug-Controlled, Multicenter, Phase III Clinical Trial. Arch Phys Med Rehabil. 2020 Sep;101(9):1485-1496. doi: 10.1016/j.apmr.2020.03.025. Epub 2020 Jun 1. PMID 32497599